CLINICAL TRIAL: NCT03057067
Title: Embolization of Pelvic Varicosities in Patients With Pelvic Congestion Syndrome
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: difficulties recruiting
Sponsor: St. Olavs Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2016/1881
Record Dates: First submitted 2017-02-15; First posted 2017-02-17 (Actual); Last update posted 2019-02-08 (Actual); Status verified 2019-02

CONDITIONS: Pelvic Pain; Varicose Veins
Keywords: Embolization, Therapeutic; Pelvis
MeSH Terms: conditions — Pelvic Pain; Varicose Veins

STUDY DESIGN:
Intervention Model Description: All female patients referred for assessment of chronic pelvic pain at the gynecological outpatient clinic or the Multidisciplinary Pain Clinic at St. Olavs Hospital are eligible for initial assessment
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- pelvic vein embolization (Experimental): female patients referred for assessment of chronic pelvic pain at the gynecological outpatient clinic or the Multidisciplinary Pain Clinic at St. Olavs Hospital, Trondheim, Norway
  Interventions: Procedure: Embolization of pelvic vein varicosities

INTERVENTIONS:
Procedure: Embolization of pelvic vein varicosities — Embolization of pelvic vein varicosities

SUMMARY:
Results of recent systematic reviews suggest favorable results of embolization for the treatment of Pelvic Congestion Syndrome (PCS) compared with pre-procedure symptoms for several outcomes, including pain reduction, overall patient satisfaction, and technical feasibility. Reported complication rates appears relatively low.

Pelvic vein embolization is a relatively new technology and the results may provide background for an evidence based decision to offer embolization of pelvic varicosities for women with PCS in Norway.

ELIGIBILITY:
Inclusion Criteria:

* Pelvic pain (lasting for more than 6 months)
* Symptoms of PCS - deterioration of pain when standing and improvement in supine position (with or without dyspareunia or dysmenorrhea).
* Confirmed pelvic varicosities by magnetic resonance examination.
* Signed, written and informed consent

Exclusion Criteria:

* Inability to communicate in Norwegian
* Known endometriosis
* Uterine myoma, uterine anomalies, or cancer
* Postmenopausal
* not having been pregnant

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 3 (Actual)
Dates: Start 2017-05-19 (Actual); Primary Completion 2019-02-07 (Actual); Study Completion 2019-02-07 (Actual)

PRIMARY OUTCOMES:
chronic pelvic pain | 3 months
  assessed by a numeric rating scale (0-10) within the questionnaire of the Norwegian Society for Pain
chronic pelvic pain | 6 months
  assessed by a numeric rating scale (0-10) within the questionnaire of the Norwegian Society for Pain
chronic pelvic pain | 1 year
  assessed by a numeric rating scale (0-10) within the questionnaire of the Norwegian Society for Pain

SECONDARY OUTCOMES:
Health related quality of life (HRQOL) | 3 months
  based on the SF-8 and mental health measurements based on the 5-mental health inventory
Health related quality of life (HRQOL) | 6 months
  based on the SF-8 and mental health measurements based on the 5-mental health inventory
Health related quality of life (HRQOL) | 1 year
  based on the SF-8 and mental health measurements based on the 5-mental health inventory
Sexual function | 3 months
  assessed with a short screening tool for sexual dysfunction, containing 4 questions plus 6 sub-questions (Hatzichristou D et al. J Sex Med 2004) - Norwegian translation (non-validated)
Sexual function | 6 months
  assessed with a short screening tool for sexual dysfunction, containing 4 questions plus 6 sub-questions (Hatzichristou D et al. J Sex Med 2004) - Norwegian translation (non-validated)
Sexual function | 1 year
  assessed with a short screening tool for sexual dysfunction, containing 4 questions plus 6 sub-questions (Hatzichristou D et al. J Sex Med 2004) - Norwegian translation (non-validated)

CONTACTS AND LOCATIONS:
Overall Officials: Risa AM Lonnee-Hoffmann, md phd, Principal Investigator — St. Olavs Hospital
Locations (1):
- St Olavs Hospital, Trondheim, Norway

IPD SHARING:
Plan to Share IPD: Undecided